CLINICAL TRIAL: NCT02435303
Title: Effect of Sildenafil for the Treatment of Sustained Pulmonary Artery Hypertension After Corrected Mitral Valve Disease
Brief Title: Effect of Sildenafil for Sustained PAH After MV Surgery (SUPERIOR Trial)
Acronym: SUPERIOR
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Number of candidates for this study is expected to be too small.
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Jong-Min Song, Professor, University of Ulsan College of Medicine, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MVsurgery_PAH
Record Dates: First submitted 2015-04-28; First posted 2015-05-06 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Hypertension, Pulmonary; Diseases of Mitral Valve
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Sildenafil (Experimental): Sildenafil 20mg tid for six months (* consider open-label extension study for 1 year)
  Interventions: Drug: Sildenafil
- Placebo (Placebo Comparator): Placebo tablets do not contain an active ingredient but are identical in shape with each active tablet of Sildenafil
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil
  Other Names: Viagra, Revatio, others
  Arms: Sildenafil
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Sildenafil is effective in the treatment of sustained pulmonary artery hypertension after corrected mitral valve disease.

ELIGIBILITY:
Inclusion Criteria:

* New York Heart Association Functional class (NYHA Fc) ≥ 2 dyspnea which was sustained till one year after the previous mitral valve surgery (repair or replacement)
* TR Vmax ≥ 3.5m/s by echocardiography
* Normal left ventricle ejection fraction (EF ≥ 50%)
* Pulmonary vascular resistance ≥ 3 Wood Unit or diastolic pressure gradient ≥ 7mmHg by cardiac catheterization

Exclusion Criteria:

* Other valve disease more than moderate degree (ex. aortic stenosis, aortic regurgitation)
* Liver cirrhosis
* Chronic renal failure with serum creatinine ≥ 1.7mg/dL
* Lung disease (ex. chronic obstructive pulmonary disease, Asthma)
* Thyroid dysfunction
* Other causes which can lead to pulmonary hypertension

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-05; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Change of Six Minutes Walk Distance | baseline and six months
  unit of measure : meter (m)

SECONDARY OUTCOMES:
Borg dyspnea score | six months
Exercise capacity by cardiopulmonary exercise test | six months
Fractional area change of right ventricle measured by echocardiography | six months
  unit of measure : percent (%)
Pulmonary vascular resistance (PVR) measured by cardiac catheterization | six months
  unit of measure : wood unit (WU)
Systolic pulmonary artery pressure measured by cardiac catheterization | six months
  unit of measure : pressure (mmHg)
Mean pulmonary artery pressure measured by cardiac catheterization | six months
  unit of measure : pressure (mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Min Song, Principal Investigator — Asan Medical Center